CLINICAL TRIAL: NCT00954083
Title: A Pilot Randomized Controlled Trial of a DIR/ Floortime Parent Training Intervention for Pre-school Children With Autistic Spectrum Disorders
Brief Title: A Pilot Trial of a Developmental, Individual-Difference, Relationship-Bases (DIR)/Floortime for Children With Autistic Spectrum Disorders
Acronym: DIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Associate Professor Dr. Kingkaew Pajareya,M.D., Rehabilitation Medicine, Siriraj Hospital, Bangkok, Thailand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 194/2550 (EC2)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Autistic Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DIR/Floortime intervention (Experimental): 1=DIR/Floortime intervention
  Interventions: Behavioral: DIR/Floortime
- routine care (Active Comparator): 2=routine care
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: DIR/Floortime — Developmental, Individual-Difference, Relationship-Bases (DIR) focus more on relationship, social skills, and meaningful, spontaneous use of language and communication and integrated understand of human development
  Arms: DIR/Floortime intervention
Behavioral: Routine care — Routine care
  Arms: routine care

SUMMARY:
Thirty two children age 2-6 years are recruited into the study and the randomization will be stratified for chronological age and symptom severity into 2 main groups, intervention and control. The intervention group will receive an additional target treatment of DIR/Floortime parent training intervention, while the control group will continue on their routine care for 3 months.

Hypothesis: Children in the intervention group show much improvement in climbing the developmental "ladder" and declining in the autistic behaviors.

ELIGIBILITY:
Inclusion Criteria:

* clinical criteria for Autistic Disorders according to DSM IV
* child is 2 - 6 years of age

Exclusion Criteria:

* children with additional medical diagnosis (e.g., genetic syndromes, diagnosed hearing impairment, diagnosed visual impairment or seizures)
* children who are geographically inaccessible for follow-up visits
* their parents are not literate or known chronic psychiatric or physical illness in the parents

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The Functional Emotional Assessment Scale (FEAS) Ratings (the child part) | at the beginning of the first session and at the 3 months follow up

SECONDARY OUTCOMES:
The Childhood Autism Rating Scale (CARS) Clinical rating of the children (6 point scale related to Greenspan's six Functional Development Level -FDL) Satisfaction of the effectiveness of the intervention of their child (Six-point Likert scale) | at the beginning of the first session and the 3 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Kingkaew Pajareya, MD, Principal Investigator — Rehabilitation Medicine, Siriraj Hospital, Bangkok, Thailand